CLINICAL TRIAL: NCT04872777
Title: Mobile Health Delivered Lifestyle Intervention Program in Patients With Nonalcoholic Steatohepatitis: A Proof of Concept Study
Brief Title: Mobile Health Delivered Lifestyle Intervention Program in Patients With NASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Noom Inc. (Industry)
Responsible Party: Principal Investigator, Jonathan Stine, Director of Research, Penn State Liver Center, Assistant Professor of Medicine and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00017544
Record Dates: First submitted 2021-04-28; First posted 2021-05-05 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Masking Description: Forty-subjects with NASH will be randomized 1:1 to either receive Noom HW mHealth lifestyle intervention or standard clinical care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Standard of care (SOC) control condition: Following study group assignment, the following procedures will be completed for SOC control:
  1. Digital scale provision (subjects may keep the scale)
  2. Reinforcement of need to comply with SOC treatment as directed by their NASH clinician
  3. Capture of available clinical information over preceding 28-days.
- Noom Healthy Weight (Experimental): Following study group assignment, the following procedures will be completed for the Noom HW mHealth lifestyle intervention:
  1. Noom application set-up and troubleshooting on smartphone (license provided)
  2. Digital scale provision (subjects may keep the scale)
  3. Capture of available clinical information over preceding 28-days.
  Interventions: Behavioral: Noom Healthy Weight

INTERVENTIONS:
Behavioral: Noom Healthy Weight — Following study group assignment, the following procedures will be completed for the Noom HW mHealth lifestyle intervention:
  1. Noom application set-up and troubleshooting on smartphone (license provided)
  2. Digital scale provision (subjects may keep the scale)
  3. Capture of available clinical information over preceding 28-days.
  Arms: Noom Healthy Weight

SUMMARY:
There is a clear unmet clinical need for effective lifestyle intervention in patients with nonalcoholic steatohepatitis (NASH). Patients have self-identified multiple barriers to effective lifestyle intervention can be removed with a mobile health (mHealth) platform.

This study will be a proof of concept study to evaluate weight loss efficacy of Noom Healthy Weight (HW), a mHealth lifestyle intervention, in patients with NASH.

ELIGIBILITY:
Inclusion Criteria:

* Adults age >18 years
* NASH defined as:
* Liver biopsy with evidence of steatohepatitis (NAS >=4) or;
* Imaging study (e.g., ultrasound, CT, MRI) with hepatic steatosis and one of the following:
* Fibroscan kPa >8.2 or;
* FAST > 0.35 or;
* FIB-4 >= 1.45 or;
* Possession of a smartphone

Exclusion Criteria:

* Active or recent (<90 days) participation in lifestyle intervention program, including weight-loss program
* Active weight-loss supplement use
* Cirrhosis
* Inability to provide informed consent
* Institutionalized/prisoner
* Other chronic liver disease (e.g., viral hepatitis)
* Recent Noom use (<180 days)
* Secondary cause of hepatic steatosis, including significant alcohol consumption (men >30g/d, women >20g/d)
* Severe medical comorbidities/psychiatric illness at the discretion of the study PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Weight | 16 weeks
  Change in self-measured body weight

SECONDARY OUTCOMES:
liver enzymes | 16 weeks
  Change in liver enzymes units per liter (alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP))
Noom healthy weight engagement | 16 weeks
  Feasibility will be assessed according to user engagement. Engaged users are defined as those who complete at least one meaningful in-application action per week (e.g., weight log, food log, exercise log, article read).
Glucose | 16 weeks
  Change in blood glucose mg/dL
hemoglobin A1c | 16 weeks
  Change hemoglobin A1c (%)
Cholesterol level | 16 weeks
  Change in cholesterol mg/dL
NAFLD Fibrosis Score | 16 weeks
  change in NAFLD Fibrosis Score
IgA level | 16 weeks
  Change in IgA level mg/dL
Ferritin | 16 weeks
  Change in Ferritin ng/mL
histology | 16 weeks
  Change in transient elastography or liver histology

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan G Stine, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Marietta, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stine JG, Rivas G, Hummer B, Duarte-Rojo A, May CN, Geyer N, Chinchilli VM, Conroy DE, Mitchell ES, McCallum M, Michealides A, Schmitz KH. Mobile health lifestyle intervention program leads to clinically significant loss of body weight in patients with NASH. Hepatol Commun. 2023 Mar 17;7(4):e0052. doi: 10.1097/HC9.0000000000000052. eCollection 2023 Apr 1. PMID 36930864